CLINICAL TRIAL: NCT02932423
Title: Impact of Beverage Consumption With Varying Sweetening Systems During Meal on Post-prandial Glucose and Insulin Concentrations, and Lipid Metabolism in Overweight and Obese Subjects
Brief Title: Metabolic Response to Beverages With Various Sweetening Systems Consumed During Meal in Overweight and Obese Subjects
Acronym: AQUAGLU-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NU377
Record Dates: First submitted 2016-10-04; First posted 2016-10-13 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Overweight and Obesity
Keywords: Sugar-sweetened beverage; Overweight; Obese; Sugar; Water
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Snack (Other): Each subject will consume 6 beverages with varying sugar content at lunch (500 ml) and with a snack in the afternoon (330 ml). The 6 beverages (Test product A, Test product B, Test product C, Test product D, Control product E and Comparative product F) will correspond to the 6 interventions.
  Interventions: Other: Control product E; Other: Test product A; Other: Test product B; Other: Test product C; Other: Test product D; Other: Comparative product F
- 2 - No snack (Other): Each subject will consume 6 beverages with varying sugar content only at lunch (500 ml). The 6 beverages (Test product A, Test product B, Test product C, Test product D, Control product E and Comparative product F) will correspond to the 6 interventions.
  Interventions: Other: Control product E; Other: Test product A; Other: Test product B; Other: Test product C; Other: Test product D; Other: Comparative product F

INTERVENTIONS:
Other: Control product E — Plain water
Other: Test product A — Beverage with no sugar but sweetener
Other: Test product B — Beverage with 22 g/L sugar and sweetener
Other: Test product C — Beverage with 33 g/L sugar and sweetener
Other: Test product D — Beverage with 47 g/L sugar and sweetener
Other: Comparative product F — Beverage with 98 g/L sugar

SUMMARY:
The purpose of this clinical study is to investigate the effect of drinking a sugar-sweetened beverage along with a meal on insulin concentrations and, glucose and lipid metabolism, in overweight and obese subjects, during a 10-hour visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject, upon briefing of the content of the present study, fully understanding and agreeing to its objective and having given written (dated and signed) informed consent form to take part in the study
* Subject who is able to communicate well with the investigator and to comply with the requirements of the entire study
* If of child bearing potential, female subject must be using or complying with one of the following medically approved methods of contraception such as, but not exclusively: oral birth control pills (at least 1 full monthly cycle prior to study product administration); intra-uterine device (IUD); double barrier methods (such as condoms and spermicide)
* Subject with a body mass index (BMI) between 25 and 35 kg/m² inclusive

Exclusion Criteria:

* Pregnant woman, based on positive urine pregnancy test, or planning to become pregnant during the study or breast-feeding woman
* Surgical operation on digestive tract, except appendectomy
* Subject who had any surgery or intervention requiring a general anaesthesia in the preceding 4 weeks, or who plans to have one during the course of the study
* Subject with diagnosed or suspected allergy or hypersensitivity to any food ingredient, including components of the study products (ingredients of sugar-sweetened beverages)
* Blood donation within the last 3 months or planning to give blood during the course of the study
* Subject involved in any other clinical study within the preceding month or in the exclusion period after another clinical study
* Subject in a situation, which in the Investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject
* Evidence of clinically relevant cardiovascular, metabolic, hematologic, hepatic, gastrointestinal, renal, pulmonary, endocrine or psychiatric history of disease as determined by medical history, physical examination, and vital signs
* Clinically significant abnormal results for urine or blood analyses

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Mean difference in maximum increment value of insulin concentration during first afternoon phase between each test product and the comparative product | 6 days (with 17 time points on each day)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne BOTTIN, PhD, Study Chair — Danone Research, Palaiseau, France
Locations (1):
- Eurofins Optimed, Gières, Auvergne-Rhône-Alpes, France